CLINICAL TRIAL: NCT02642523
Title: Natriuretic Peptides and Metabolic Risk in Obesity
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Preliminary data run on rat samples showed that this study question and design would not produce conclusive results. The PI decided not to carry out the study.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Thomas Wang, Principal Investigator, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 151768
Record Dates: First submitted 2015-11-24; First posted 2015-12-30 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Hyperinsulinemia
Keywords: natriuretic peptide; insulin; lipolysis; hormones; metabolism
MeSH Terms: conditions — Obesity; Hyperinsulinism; Insulin Resistance | interventions — Natriuretic Peptide, Brain; Insulin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saline Infusion (Placebo Comparator): All subjects will undergo 3 interventions, performed at 3 separate outpatient study visits. The order of the 3 interventions will be randomly assigned. The interventions are: Saline Infusion, Insulin Clamp, and BNP Infusion (Nesiritide).
  Interventions: Other: Saline
- Insulin Clamp (Experimental): All subjects will undergo 3 interventions, performed at 3 separate outpatient study visits. The order of the 3 interventions will be randomly assigned. The interventions are: Saline Infusion, Insulin Clamp, and BNP Infusion (Nesiritide).
  Interventions: Drug: Insulin
- BNP Infusion (Nesiritide) (Experimental): All subjects will undergo 3 interventions, performed at 3 separate outpatient study visits. The order of the 3 interventions will be randomly assigned. The interventions are: Saline Infusion, Insulin Clamp, and BNP Infusion (Nesiritide).
  Interventions: Drug: Nesiritide

INTERVENTIONS:
Drug: Nesiritide — Subjects will receive an intravenous infusion of recombinant human b-type natriuretic peptide (BNP) (Nesiritide) over 2 hours at 2 doses: 0.003 ug/kg/min for 1 hour, followed by 0.01 ug/kg/min for 1 hour. Nesiritide (Johnson and Johnson) is FDA-approved for the treatment of heart failure. Study investigators received approval from the FDA for an IND exemption for nesiritide in this study. While receiving the BNP infusion, subjects will also receive an intravenous infusion of normal (0.9%) saline over 2 hours. Subjects will receive a standardized high-salt diet for at least 6 days prior to this study visit.
  Other Names: Recombinant human BNP
  Arms: BNP Infusion (Nesiritide)
Drug: Insulin — The hyperinsulinemic-euglycemic insulin clamp, which will last between 2-2.5 hours, involves continuous intravenous infusions of human regular insulin and of dextrose solution. Simultaneously, subjects receive an intravenous infusion of normal (0.9%) saline over 2 hours. Subjects will receive a standardized high-salt diet for at least 6 days prior to this study visit.
  Other Names: Human Insulin
  Arms: Insulin Clamp
Other: Saline — Subjects will receive an intravenous infusion of normal (0.9%) saline over 2 hours at a rate of 0.25 ml/kg/min. Subjects will receive a standardized high-salt diet for at least 6 days prior to this study visit.
  Other Names: Normal Saline
  Arms: Saline Infusion

SUMMARY:
The investigators are examining:

1. the relationships of insulin levels and natriuretic peptide hormone levels, and
2. the effects of administering an infusion of natriuretic peptide hormone on the breakdown of fat

in healthy lean and otherwise healthy obese individuals.

DETAILED DESCRIPTION:
The cardiac natriuretic peptide hormonal system may protect against the development of cardiometabolic risk. Epidemiologic studies have shown that in relatively healthy individuals without heart failure, low natriuretic peptide levels are associated with unfavorable cardiometabolic phenotypes, including higher blood pressure, obesity, higher insulin levels, and diabetes mellitus. Understanding the mechanisms behind the "natriuretic peptide deficiency" of obesity would illuminate an important way in which obesity interacts with the cardiovascular system.

The investigators propose a prospective cross-over design in 40 healthy lean and otherwise healthy obese individuals. The investigators propose the following specific aims and hypotheses:

Aim 1: To study the effect of hyperinsulinemia on the response of the natriuretic peptide system to salt loading.

Hypothesis 1: Hyperinsulinemia will suppress natriuretic peptide levels in both obese and lean individuals.

Aim 2: To examine the effect of an intravenous infusion of natriuretic peptide on acute markers of lipolysis.

Hypothesis 2: An intravenous infusion of natriuretic peptide will raise acute markers of lipolysis in both obese and lean individuals.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-50 years
* BMI 18 to <25 kg/m2 (lean group, N=20) or BMI 30 to <40 kg/m2 (obese group, N=20)

Exclusion Criteria:

* Current use of antihypertensive medications
* Current use of glucocorticoids, metformin, or any antidiabetes medications
* Prior or current cardiovascular disease, renal disease, or liver disease
* Diabetes mellitus (taking insulin, other anti-diabetic agents, or diet-controlled)
* Atrial fibrillation
* Bleeding disorder or anemia
* Elevated LFTs
* estimuated GFR < 60 ml/min
* Abnormal sodium or potassium level
* Positive pregnancy test, women of child-bearing age not practicing birth control, women who are breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in natriuretic peptide levels | 4 hours (during 2-hour study infusions and for 2 hours after study infusions)
Change in glycerol levels | 1 hour
  Change during 1-hour of low-dose BNP infusion, 1-hour of high-dose BNP infusion, and 1-hour of normal saline infusion

SECONDARY OUTCOMES:
Change in free fatty acid levels | 1 hour
  Change during 1-hour of low-dose BNP infusion, 1-hour of high-dose BNP infusion, and 1-hour of normal saline infusion
Change in triglyceride levels | 1 hour
  Change during 1-hour of low-dose BNP infusion, 1-hour of high-dose BNP infusion, and 1-hour of normal saline infusion
Change in energy expenditure assessed by indirect calorimetry | 1 hour
  Change during 1-hour of low-dose BNP infusion, 1-hour of high-dose BNP infusion, and 1-hour of normal saline infusion

OTHER OUTCOMES:
Change in plasma renin activity | 4 hours (during 2-hour study infusions and for 2 hours after study infusions)
Change in aldosterone | 4 hours (during 2-hour study infusions and for 2 hours after study infusions)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine N Bachmann, MD, Study Director — Vanderbilt Diabetes/Endocrinology; Thomas J Wang, MD, Principal Investigator — Vanderbilt Cardiovascular Medicine